CLINICAL TRIAL: NCT06261151
Title: Preoperative Nutritional Status and Risk Factors Associated With Delayed Discharge in Elderly Patients Undergoing Gastrectomy: A Single-center Retrospective Study
Brief Title: Preoperative Nutritional Status Associated With Delayed Discharge in Elderly Patients Undergoing Gastrectomy
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Zhongshan-HHY-03
Record Dates: First submitted 2024-02-08; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Preoperative Nutritional Status and Risk Factors Associated With Elderly Patients Undergoing Gastrectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Clinical data collection — Clinical data of elderly patients with gastric cancer who underwent open gastrectomy were collected and analyzed.

SUMMARY:
Gastric cancer (GC) remains the 5th most common cancer worldwide and had the second- highest mortality rate in China. The population of elder patients with GC has been increasing because of the high prevalence of H. pylori infection and increasing life expectancy. Elderly GC patients face several challenges during treatment, such as comorbidities, organ dysfunction, immunosuppression, and delayed recovery. Advanced age is associated with a higher rate of postoperative complications shortly after surgical treatment, and lower 5-year overall survival as long-term outcome.

In China, the prevalence of malnutrition in hospitalized patients is around 12.6% to 46.19%. Malnutrition is one of the great risk factors of adverse clinical outcomes in elderly patients with GC. The nutritional status at the time of diagnosis was independently associated with postoperative complications, overall survival, and disease-free survival. The condition can be caused by mechanical obstruction of the digestive tract or anorexia-cachexia syndrome, leading to insufficient protein or energy intake and absorption disorder. Nutrition screening, assessment, and intervention are important steps in nutritional management.

Previous studies mostly focused on hospitalized internal medical patients. Only a few studies focused on surgical patients regardless of age. Therefore, in this retrospective study, we are going to investigate the nutritional status and perioperative nutritional support of geriatric surgical patients with GC, and provide a basis for implementing an effective nutritional intervention.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 60-90 years old; Patients with gastric cancer; Patients who underwent radical gastrectomy. -

Exclusion Criteria:

Patients with other malignancies; Patients with previous gastrointestinal surgery or emergency surgery; Patients with incomplete medical record.

-

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 60-90 years old with gastric cancer who underwent radical gastrectomy were retrospectively analyzed from the prospectively collected database of Zhongshan Hospital of Fudan University between March 2024 and December 2024.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
The preoperative nutritional status of elderly patients underwent gastrectomy | March 01, 2024 to December 31, 2024.
  According to the European Society for Clinical Nutrition and Metabolism (ESPEN) diagnostic criteria, malnutrition is defined as a weight loss of more than 10% (indefinite of time) or more than 5% over the last 3 months and a body mass index (BMI)<20 kg/m2 or <22 kg/m2 in patients under or above the age of 70, respectively. Nutritional assessment is performed based on a prognostic nutritional index (PNI), which is calculated based on the equation: [(10×serum albumin (g/dL)) + (0.005×total lymphocyte count (/mm3))].